CLINICAL TRIAL: NCT04844671
Title: Patients' Expectations About Effects of Robotic Surgery for Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2021LSK-068
Record Dates: First submitted 2021-04-04; First posted 2021-04-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cancer; Robotic Surgery; Patients' Expectations
Keywords: Patients' Expectations; Robotic surgery; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: da Vinci Surgical Systems — The da Vinci Surgical Systems enable surgeons to perform delicate and complex operations through a few small incisions with robotic assisted surgery.

SUMMARY:
Robotic surgery for common surgical procedures is on the rise despite limited evidence to support its clinical benefit. We intend to to map and characterize the prevalence of the patients'expectation that robotic surgery might be superior to open or laparoscopic procedures and to identify the sociodemographic, clinical and organisational factors associated with this expectation.

DETAILED DESCRIPTION:
With the progress of modern medicine, minimally invasive surgical technology has become the main theme in the field of contemporary surgery. As a rising star, the Da Vinci robotic surgery system provides surgeons with a more comprehensive surgical vision, more flexible instrument control, finer anatomy, and more natural comfort compared to open surgery and laparoscopic surgery. However, due to the lack of long-term theoretical basis, the evidence to support its clinical benefits is limited, and its application is limited by related postoperative complications and high operation-related costs. At present, the number of Da Vinci robotic surgery is steadily increasing around the world, but what are the expectations of patients that robotic surgery may be better than open or laparoscopic surgery? It is also unclear what reasons are related to this established expectation. Therefore, we intend to map and characterize the prevalence of the patients' expectation that robotic surgery might be superior to open or laparoscopic procedures and to identify the sociodemographic, clinical and organisational factors associated with this expectation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cancer
* Have undergone tumor resection with Da Vinci Robotic Surgery System
* Volunteer to participate in the study

Exclusion Criteria:

* Patients with mental illness
* Cognitive dysfunction
* Cannot complete the questionnaire independently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone Da Vinci robotic surgery in the first affiliated hospital of Xi'an Jiaotong University in the past five years
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Factors Associated With Patients' Decisions Factors Associated With Patients'Decisions to Choose Robotic Surgery | 2021.4-2022.4
  Factors Associated With Patients'Trends in the Adoption of Robotic Surgery for Common Surgical Procedures。According to the relevant regulations of the hospital inpatient satisfaction survey, we have developed a satisfaction rating scale, the evaluation is divided into five grades: "very satisfied" = 5, "relatively satisfied" = 4, "general" = 3, "not very satisfied" = 2, "very dissatisfied" = 1, the total score is 1-5.

SECONDARY OUTCOMES:
Social demographic characteristics | 2021.4-2022.4
  Age, Sex, Education, Occupation
Economic status | 2021.4-2022.4
  The ability to pay for medical expenses and the type of medical insurance.Based on the types of medical insurance in China, our survey design is divided into four categories: 1. China new rural cooperative medical system; 2. The medical insurance for urban residents; 3. The medical insurance for urban workers; 4. Commercial insurance. According to China's national income level, our survey design is divided into three stages: personal annual income below 50,000 RMB, 50,000-100,000 RMB, and more than 100,000 RMB.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhang, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol